CLINICAL TRIAL: NCT01163071
Title: A Phase I Trial of ABI-011 Administered Weekly in Patients With Advanced Solid Tumors or Lymphomas
Brief Title: A Phase 1 Trial of ABI-011 in Patients With Advanced Solid Tumors or Lymphomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA601
Record Dates: First submitted 2010-06-15; First posted 2010-07-15 (Estimated); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABI-011 (Experimental)
  Interventions: Drug: ABI-011

INTERVENTIONS:
Drug: ABI-011 — ABI-011

SUMMARY:
The purpose of this study is to determine the MTD and/or RP2D of ABI-011 when administered by IV on Day 1, Day 8 and Day 15 with one week of rest for patients with advanced solid tumor malignancies and lymphomas.

DETAILED DESCRIPTION:
Dose limiting toxicities (DLT), maximum tolerated dose (MTD)

ELIGIBILITY:
Inclusion Criteria:

* Must be equal or greater 18 years of age
* ECOG performance status less than or equal to 2 (Appendix 2)
* Pts. must be willing and able to sign informed consent
* Cytologically or histologically confirmed solid tumor malignancy or lymphoma for which no standard approved therapy is available. Patients should have accessible tumor lesions amendable to 2 serial biopsies which would not put the patient or their treatment at risk
* Pt. agrees and is willing to provide 2 serial tumor biopsies(optional on first phase, mandatory on 2nd phase)
* During the dose escalation phase, measurable or non-measurable disease as defined by RECIST criteria. At 2nd phase, only patients with measurable disease
* Life expectancy of equal or greater than 12 weeks
* All AEs of any prior chemotherapy, surgery or radiotherapy, must have resolved to grade equal to or less than 1
* The following laboratory results must be present within 14 days of initial ABI-011 administration

  * Hemoglobin greater or equal to 9g/dL
  * Absolute neutrophils count(ANC)greater or equal to 1.5 x 10^9/L
  * Platelet count is greater or equal to 100 x 10^9/L
  * Serum bilirubin less than or equal to 1.5 x upper limit of normal (ULN)
  * Aspartate transaminase (AST) and alanine transaminase (ALT)is less than or equal to 2.5 ULN(except if liver metastases are present; then values must be less than or equal to 5 x ULN)
  * Potassium, corrected calcium and magnesium WNL
  * Serum Creatinine less than or equal to 1.5 x ULN
  * Activated aPTT,PT,INR,WNL
  * WNL levels : Troponin I and T, CK-MB,BNP
* At least one measurable lesion should be evaluable (DCE-MRI eligibility criteria)and meet at least one of the criteria below:

  * At least one measurable lesions should be at least 3 cm in diameter and should not be near the diaphragm or mediastinum
  * Lesions should be solid masses that enhance with contrast, without signs of calcification on the most recent computed tomography (CT) or magnetic resonance (MRI)scan
* Pts. must be willing to practice contraceptive methods for the duration of the study and for one month following study completion. Female patients must be postmenopausal, surgically sterile or they must agree to use acceptable methods of birth control. Male patients must be surgically sterile or agree to use an acceptable method of contraception.
* Women of childbearing potential must have a negative serum pregnancy test(B-hCG)within 72 hours prior to first study drug administration

Exclusion Criteria:

* Inability to comply with study and follow-up procedures
* Women who are pregnant or lactating
* Treatment with chemotherapy, hormonal therapy(except leuprolide for prostate cancer), immunotherapy, biologic therapy, or radiation therapy as cancer therapy within 4 weeks before initiation of study treatment. Six weeks should have elapsed if prior chemotherapy treatment included nitrosoureas or mitomycin C
* Pts. who have received antibody-based therapies within 28 days or 5 half-lives of the agent, whichever time period is longer
* Major surgery within 6 weeks before first study drug administration
* Prior treatment with tumor vascular disruptive agents
* Any uncontrolled medical or psychiatric risk factors
* Central nervous system(CNS)metastases.
* History of diabetic retinopathy. All patients must be evaluated by an ophthalmologist prior to study treatment
* Any history of myopathy, either peripheral or cardiac
* Current use of medications that may have the potential of QTc prolongation
* History of allergy or hypersensitivity to any compound of the ABI-011 formulation
* Active uncontrolled bacterial, viral, or fungal infection, requiring systemic therapy
* Pt.has known infection with human immunodeficiency virus (HIV),or known chronic Hepatitis B or Hepatitis C
* Inability to be venipunctured and/or tolerate venous access
* History of other carcinoma within past 5 years
* Pts. requiring therapeutic anticoagulation with either coumadin or low molecular weight heparin or with history of any bleeding diathesis. Low dose aspirin and low dose coumadin for catheter maintenance are allowed
* Lung tumors in a central position.
* Cardiac exclusion criteria:

  * Left ventricular ejection fraction (LVEF)< 50% by echocardiography;
  * Previous history of MI or ischemic heart disease
  * EKG findings suggestive of current or previous ischemic heart disease, including left bundle branch block
  * Prior treatment with chemotherapy agents known to potentially cause cardiotoxicity
  * Class III or IV heart failure as defined by the New York Heart(NYHA) functional classification
  * Congenital or acquired long QT syndrome
  * Uncontrolled hypertension
  * Current or past history of clinically significant arrhythmias
  * QTc prolongation
  * HO Symptomatic PVD (Venous or arterial)
* Seizure disease requiring current anticonvulsant treatment
* HO previous CVA or TIA
* HO inflammatory bowel disease (active or past) or active PUD
* HO previous, whole abdomen radiation therapy or more than Grade 1 residual toxicity from previous radiation therapy.
* History of autoimmune disease or vascular disease (venous or arterial)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-03-01 (Actual); Primary Completion 2011-09-23 (Actual); Study Completion 2011-09-23 (Actual)

PRIMARY OUTCOMES:
DLT's and MTD Safety and Toxicity profile | During Cycle 1, treatment period, End of Study and Follow-Up, approximately up to 2 years
  Evaluate PK and PD of ABI-011. Preliminary assessment of tumor response.

SECONDARY OUTCOMES:
Safety and toxicity profile of repeated dosing of ABI-011 | End of study and follow up, approximately up to 2 years
  Number of subjects with Adverse Events; laboratory assessments, ECG assessments, opthalmologic assessments
Evaluate plasma PK of ABI-011 on this schedule | End of Study and follow-up, Up to two years
Assess biological activity and PD of ABI-011 | End of study and follow-up, approximately 2 years
Make preliminary assessment of tumor response | End of study and follow-up, approximately 2 years
Assess biological activity/exploratory during treatment C1, C2, EOS | End of Study and follow-up, aproximately two years

CONTACTS AND LOCATIONS:
Overall Officials: Patricia M LoRusso, DO, Principal Investigator — Karmanos Cancer Institute Hudson-Webber Cancer Research Center; John Sarantopoulos, MD, Principal Investigator — Cancer Therapy Research Center at the University Health Sciences Center at San Antonio
Locations (2):
- United States (2):
  - Karmanos Cancer Center Institute, Detroit, Michigan
  - CTRC @ The Utah Health Science Center @ San Antonio, San Antonio, Texas